CLINICAL TRIAL: NCT03717428
Title: Preventing Age-Related Weight Gain in the Workplace With Daily Weighing
Acronym: Weigh2Go
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1606006401
Record Dates: First submitted 2018-05-17; First posted 2018-10-24 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Effect of self-weighing to prevent age-related weight gain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Weighing Group (Experimental): This group will be weighed and height measured in our metabolic unit at the beginning and end of the two year experimental period. In addition, the intervention in Daily Weighing Group is that they will be given an internet based scale and asked to weigh themselves immediately after rising from bed every morning for the duration of the two year experimental period.
  Interventions: Device: Daily Weighing Group
- Control Group (Active Comparator): The only intervention for the control group is that they will be weighed and height measured at the beginning and end of the experimental period in our metabolic unit.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Daily Weighing Group — The Experimental group will weigh themselves everyday
  Other Names: Daily weighing
  Arms: Daily Weighing Group
Device: Control group — This group will be weighed and measured at the beginning and end of the study and will not be weighing themselves daily
  Other Names: Not weighing daily
  Arms: Control Group

SUMMARY:
To examine the effectiveness of daily weighing to prevent age-related weight gain.

DETAILED DESCRIPTION:
Cornell employee's were recruited for a two-year weight gain prevention study. Height and weights were taken in our metabolic center. They were randomized into two group. The experimental group was given an internet based scale and asked to weigh themselves every morning immediately after rising. The other group was asked to return at the end of the study when they height and weight will again be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-diabetic

Exclusion Criteria:

* History of eating disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Weight Change | 2 year
  body weight

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stover, Study Director — Cornell University

IPD SHARING:
Plan to Share IPD: No